CLINICAL TRIAL: NCT07321860
Title: Randomized, Double-Blind, Placebo-Controlled Phase 2a Study of Partial TGF-βR1 (ALK5) Inhibition With Galunisertib Combined With PDE4 Inhibition With Nerandomilast in GREM2-Positive ALS
Brief Title: This Study Evaluates the Safety, Target Engagement, and Preliminary Efficacy of Galunisertib (TGF-βR1/ALK5 Inhibitor)Combined With Nerandomilast (PDE4 Inhibitor) in GREM2-positive ALS, a Biomarker-defined Subgroup Hypothesized to Reflect Heightened TGF-β/SMAD-driven Astrocytic and Fibrotic Signaling
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gipfel Life Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GALNERAN-KI
Record Dates: First submitted 2026-01-02; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — LY-2157299

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Galunisertib + Nerandomilast Combination (Active Comparator)
  Interventions: Drug: Galunisertib + Nerandomilast Combination
- Placebo (Placebo Comparator)
  Interventions: Drug: Galunisertib + Nerandomilast Combination

INTERVENTIONS:
Drug: Galunisertib + Nerandomilast Combination — Galunisertib + Nerandomilast Combination

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a relentlessly progressive neurodegenerative disorder characterized by loss of upper and lower motor neurons, leading to muscle weakness, respiratory decline, and eventual mortality. A growing body of translational and clinical evidence implicates neuroinflammation, reactive astrocytosis, and maladaptive TGF-β signaling as central contributors to disease progression. Elevated levels of Gremlin-2 (GREM2) have been identified as a marker of dysregulated TGF-β-linked astrocytic activity and fibrotic gene programs in some ALS patients, and preclinical data suggest that attenuating these pathways may mitigate glial toxicity and improve neuronal survival.

Galunisertib, a selective ATP-competitive TGF-β receptor type I (TGF-βR1/ALK5) inhibitor, has been developed to block SMAD2/3 phosphorylation and TGF-β-mediated transcriptional programs. Meanwhile, nerandomilast, a selective PDE4B inhibitor, elevates intracellular cAMP in immune and glial cells, shifting pro-inflammatory signaling toward resolution and antagonizing secondary fibrotic and inflammatory cascades. Preclinical models show that PDE4 inhibition and TGF-β pathway blockade concurrently reduce maladaptive glial phenotypes and fibrotic mediators.

This study investigates the combination of galunisertib + nerandomilast in ALS patients with elevated GREM2, hypothesizing that dual targeting of TGF-β-mediated astrocytic reactivity and PDE4B-regulated inflammatory signaling will translate into slowing of disease progression and favorable pharmacodynamic effects on central biomarkers of neuroinflammation and neurodegeneration.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

1. Age:

   * 18 to 80 years, inclusive, at the time of informed consent.
2. Diagnosis of ALS:

   * Diagnosis of amyotrophic lateral sclerosis according to revised El Escorial criteria or equivalent, confirmed by a qualified neurologist.
3. GREM2-Positive Status:

   * Evidence of elevated GREM2 at screening, defined as:
   * CSF GREM2 above a pre-specified threshold OR
   * Plasma GREM2 above a pre-specified threshold with supportive evidence of astrocytic or TGF-β pathway activation (e.g., elevated GFAP or TGF-β-responsive biomarker).
   * Biomarker thresholds will be defined prospectively in the protocol and laboratory manual.
4. Disease Duration:

   * Time from first ALS-related symptom onset ≤ 24 months at screening.
5. Functional Status:

   * ALS Functional Rating Scale - Revised (ALSFRS-R) total score ≥ a protocol-defined minimum (e.g., ≥ 25) at screening, sufficient to allow detection of functional change.
6. Respiratory Function:

   * Slow vital capacity (SVC) or forced vital capacity (FVC) ≥ 50% of predicted at screening.
7. Stable Background ALS Therapy:

   * If receiving riluzole and/or edaravone, participants must be on a stable dose for ≥ 30 days prior to screening and willing to maintain the regimen throughout the study.
8. Ability to Consent:

   * Ability to understand and provide written informed consent personally or via a legally authorized representative, in accordance with local regulations.
9. Contraception:

   * Women of childbearing potential and men with partners of childbearing potential must agree to use effective contraception during the study and for a defined period after the last dose.

Exclusion Criteria

Participants will be excluded if any of the following apply:

1. Non-ALS Motor Neuron Disease:

   * Diagnosis of primary lateral sclerosis (PLS), progressive muscular atrophy (PMA), or other non-ALS motor neuron disorders.
2. Advanced Respiratory Insufficiency:

   * Requirement for invasive mechanical ventilation at screening or anticipated need within the immediate study period.
3. Clinically Significant Hepatic Disease:

   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN) at screening.
   * Known cirrhosis or active chronic liver disease.
4. Clinically Significant Cardiac Disease:

   * Uncontrolled arrhythmia, recent myocardial infarction, unstable angina, or clinically significant cardiac dysfunction that may increase risk with study participation.
5. Active or Uncontrolled Infection:

   * Active systemic infection requiring treatment at screening or known chronic infection that could interfere with immune or biomarker assessments.
6. Immunocompromised State:

   * History of organ transplantation, active malignancy requiring systemic therapy, or chronic immunosuppressive therapy (excluding stable low-dose corticosteroids, if allowed by protocol).
7. Prior Exposure to TGF-β Pathway Inhibitors:

   * Previous treatment with galunisertib or other direct TGF-β or ALK5 inhibitors within a protocol-defined washout period.
8. Recent Investigational Therapy:

   * Participation in another interventional clinical trial or receipt of an investigational drug within 30-60 days prior to screening (exact window defined in protocol).
9. Concomitant Medications with High Interaction Risk:

   * Use of strong CYP modulators or medications known to significantly interfere with galunisertib or nerandomilast metabolism, unless safely discontinued.
10. Pregnancy or Breastfeeding:

    * Pregnant or breastfeeding women.
11. Other Medical Conditions:

    * Any medical, neurological, or psychiatric condition that, in the investigator's judgment, could:
    * Interfere with study participation or compliance,
    * Confound interpretation of efficacy or biomarker outcomes,
    * Increase risk to the participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic Biomarkers - Change from Baseline in GREM2 and TGF-β Pathway Marker Levels | Time Frame: Baseline to 24 Weeks
  Pharmacodynamic Biomarkers - Change from Baseline in GREM2 and TGF-β Pathway Marker Levels (CSF or plasma; Time Frame: Baseline to 24 Weeks). Definition: GREM2 (Gremlin-2) concentration in cerebrospinal fluid or plasma will be measured at baseline and 24 weeks. GREM2 is a TGF-β-inducible protein ￼ used to stratify patients (GREM2-positive) and serves as a proxy for TGF-β pathway activity. In addition, downstream TGF-β signaling biomarkers will be assessed over the same period, including phosphorylated SMAD2/3 (pSMAD2/3) in peripheral blood cells and plasminogen activator inhibitor-1 (PAI-1, SERPINE1) in plasma. These are direct readouts of TGF-β receptor activity ￼ and are strongly upregulated by TGF-β signaling ￼. Glial/neuroinflammatory markers such as glial fibrillary acidic protein (GFAP) and neurofilament light chain (NfL) in CSF or blood will also be measured, as they indicate astrocyte activation and neuroaxonal injury in ALS ￼. Analysis: Changes from baseline in GREM2 and the